CLINICAL TRIAL: NCT04017663
Title: Publicly Versus Privately-Funded Cardiac Rehabilitation: Access and Adherence Barriers
Brief Title: Publicly Versus Privately-Funded Cardiac Rehabilitation
Status: Completed | Type: Observational
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mayara Moura Alves da Cruz, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Other Study IDs: CAAE: 88504718.0.0000.5402
Record Dates: First submitted 2019-07-04; First posted 2019-07-12 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: Rehabilitation; Surveys and Questionnaires; Treatment Adherence and Compliance; Patient Compliance
MeSH Terms: conditions — Cardiovascular Diseases; Treatment Adherence and Compliance; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Public group: patients who performed cardiovascular rehabilitation in a public center
  Interventions: Other: Application of questionnaires
- Private group: patients who performed cardiovascular rehabilitation in a private center
  Interventions: Other: Application of questionnaires

INTERVENTIONS:
Other: Application of questionnaires — Application of questionnaires to identify characteristics and main barriers of patients

SUMMARY:
This is an observational cross-sectional study designed to investigate the barriers encountered by patients after admission to a public and private PRC and to correlate the barriers with the population profile.

To participate in this study, patients were recruited for convenience of two CRPs offered in the city of Presidente Prudente - SP, one linked to the private service offered by the Heart Institute (INCOR) and another public in the Cardiology Sector of the Center for Studies and Attendance in Physiotherapy and Rehabilitation - CEAFiR of the Faculty of Sciences and Technology, State University of São Paulo, Júlio de Mesquita Filho (FCT-UNESP).

As eligibility criteria, patients over 18 years of age, regardless of sex, diagnosed with cardiovascular diseases or referred for risk factor prevention and who had attended CRP for at least 3 months, regardless of the frequency percentage, were considered. Patients who were not found after three visits to the programs for evaluation were excluded from the study.

After the initial invitation and evaluation of the eligibility criteria, the participants were informed about the procedures and objectives of the study, and after agreeing, they signed the informed consent form. The study protocol was approved by the Research Ethics Committee of FCT-UNESP under CAAE number: 88504718.0.0000.5402.

For this, in only one meeting, an initial evaluation was made in order to identify and characterize the patients. Four questionnaires were then applied: the Brazilian Association of Research Companies (ABEP) Questionnaire for the evaluation of socioeconomic level, Mini Mental State Examination (MMSE), Hospital Anxiety and Depression Scale (HADS) and Barrier Scale for Cardiac Rehabilitation (EBRC).

Barriers were considered as the primary end point and correlations with the population profile as secondary outcomes.

DETAILED DESCRIPTION:
This is an observational cross-sectional study designed to investigate the barriers encountered by patients after admission to a public and private PRC and to correlate the barriers with the population profile.

To participate in this study, patients were recruited for convenience of two CRPs offered in the city of Presidente Prudente - SP, one linked to the private service offered by the Heart Institute (INCOR) and another public in the Cardiology Sector of the Center for Studies and Attendance in Physiotherapy and Rehabilitation - CEAFiR of the Faculty of Sciences and Technology, State University of São Paulo, Júlio de Mesquita Filho (FCT-UNESP).

As eligibility criteria, patients over 18 years of age, regardless of sex, diagnosed with cardiovascular diseases or referred for risk factor prevention and who had attended CRP for at least 3 months, regardless of the frequency percentage, were considered. Patients who were not found after three visits to the programs for evaluation were excluded from the study.

After the initial invitation and evaluation of the eligibility criteria, the participants were informed about the procedures and objectives of the study, and after agreeing, they signed the informed consent form. The study protocol was approved by the Research Ethics Committee of FCT-UNESP under CAAE number: 88504718.0.0000.5402.

For this, in only one meeting, an initial evaluation was made in order to identify and characterize the patients. Four questionnaires were then applied: the Brazilian Association of Research Companies (ABEP) Questionnaire for the evaluation of socioeconomic level, Mini Mental State Examination (MMSE), Hospital Anxiety and Depression Scale (HADS) and Barrier Scale for Cardiac Rehabilitation (EBRC).

Regarding the initial evaluation, the patients were asked about their age, weight and height to obtain the body mass index (BMI) 23, occupation, schooling, city where they currently reside, clinical diagnosis and time of rehabilitation treatment.

In addition, socioeconomic level, cognitive status and level of anxiety and depression were evaluated, which together with the information obtained in the initial evaluation provided the population profile.

In relation to the questionnaires, the questionnaire of the Brazilian Association of Companies and Research (ABEP) was used to analyze the socioeconomic level, which includes the level of schooling, and includes questions about family income, possession of public items and services offered in its residence. The sum of the points can result in a value between zero and one hundred points and the higher the score obtained in the questionnaire the greater the economic power of the patient. From the obtained score, the questionnaire allows the classification of the individual in classes A (average family income of R $ 20,888), B1 (average family income of R $ 9,254), B2 (average family income of R $ 4,852), C1 average family income of R $ 2,705), C2 (average family income of R $ 1,625), D and E (average family income of R $ 3,130), with A for a score higher than 45 and E, a score lower than 16.

The Mental State Mini Exam (MMSE) was used to assess cognitive status. The test is subdivided into two sections, the first one evaluates the orientation, memory and attention and in the second, the ability to appoint, from obedience to a verbal and written command, free writing of a sentence and copy of a complex drawing ( polygons). The higher the score obtained in the test, the better the patient's cognitive status, also considering the level of education (cutoff points: 20 points for illiterates, 25 points for individuals with 1 to 4 years of study, 26.5 points for individuals with 5 to 8 years of study, 28 points for individuals with 9 to 11 years of study, 29 points for individuals with more than 11 years of study).

To quantify the level of anxiety and depression, the Hospital Anxiety and Depression Scale (HADS) was applied. This scale presents seven affirmations for classifying anxiety and seven for depression, which present four options of responses ranging from zero to three points, which generates two scores, one for anxiety and another for depression. The classification is distributed between unlikely anxiety disorder or depression (0 to 7 points), possible disorder (8 to 11 points) and probable disorder (12 to 21 points).

Barriers were evaluated through the Barrier Scale for Cardiac Rehabilitation (EBRC), which is composed of twenty-one items that are scored using a Likert scale, which varies from one to five. This scale can be analyzed by the mean score of all items or divided into five subscales: comorbidities / functional status (B1: items 8, 9, 13, 14, 15, 17 and 21), perceived needs (B2: items 3 (B3: items 4, 7 and 18), travel / work conflicts (B4: items 10 and 12) and access (B5: items 1, 2, 19 and 20) 13. The higher the result of the averages, the greater the number of barriers found.

Barriers were considered as the primary end point and correlations with the population profile as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* As eligibility criteria, patients over 18 years of age, regardless of sex, diagnosed with cardiovascular diseases or referred for risk factor prevention and who had attended CRP for at least 3 months, regardless of the frequency percentage, were considered.

Exclusion Criteria:

* Patients who were not found after three visits to the programs for evaluation were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To participate in this study, patients were recruited for convenience of two CRPs offered in the city of Presidente Prudente - SP, one linked to the private service offered by the Heart Institute (INCOR) and another public in the Cardiology Sector of the Center for Studies and Attendance in Physiotherapy and Rehabilitation - CEAFiR of the Faculty of Sciences and Technology, State University of São Paulo, Júlio de Mesquita Filho (FCT-UNESP).
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Barriers | In the first 1 day of avaliation
  Barriers were evaluated through the Barrier Scale for Cardiac Rehabilitation (EBRC), which is composed of twenty-one items that are scored using a Likert scale, which varies from one to five. This scale can be analyzed by the mean score of all items or divided into five subscales: comorbidities / functional status (B1: items 8, 9, 13, 14, 15, 17 and 21), perceived needs (B2: items 3 (B3: items 4, 7 and 18), travel / work conflicts (B4: items 10 and 12) and access (B5: items 1, 2, 19 and 20) 13. The higher the result of the averages, the greater the number of barriers found.
Socieconomic level | In the first 1 day of avaliation
  In relation to the questionnaires, the questionnaire of the Brazilian Association of Companies and Research (ABEP) was used to analyze the socioeconomic level, which includes the level of schooling, and includes questions about family income, possession of public items and services offered in its residence. The sum of the points can result in a value between zero and one hundred points and the higher the score obtained in the questionnaire the greater the economic power of the patient. From the obtained score, the questionnaire allows the classification of the individual in classes A (average family income of R $ 20,888), B1 (average family income of R $ 9,254), B2 (average family income of R $ 4,852), C1 average family income of R $ 2,705), C2 (average family income of R $ 1,625), D and E (average family income of R $ 3,130), with A for a score higher than 45 and E, a score lower than 16.
Cognitive Status | In the first 1 day of avaliation
  The Mental State Mini Exam (MMSE) was used to assess cognitive status. The test is subdivided into two sections, the first one evaluates the orientation, memory and attention and in the second, the ability to appoint, from obedience to a verbal and written command, free writing of a sentence and copy of a complex drawing ( polygons). The higher the score obtained in the test, the better the patient's cognitive status, also considering the level of education (cutoff points: 20 points for illiterates, 25 points for individuals with 1 to 4 years of study, 26.5 points for individuals with 5 to 8 years of study, 28 points for individuals with 9 to 11 years of study, 29 points for individuals with more than 11 years of study).
Anxiety and depression level | In the first 1 day of avaliation
  To quantify the level of anxiety and depression, the Hospital Anxiety and Depression Scale (HADS) was applied. This scale presents seven affirmations for classifying anxiety and seven for depression, which present four options of responses ranging from zero to three points, which generates two scores, one for anxiety and another for depression. The classification is distributed between unlikely anxiety disorder or depression (0 to 7 points), possible disorder (8 to 11 points) and probable disorder (12 to 21 points).

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna LB Borges, Principal Investigator — São Paulo State University (UNESP)
Locations (1):
- Unesp, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No